CLINICAL TRIAL: NCT06208202
Title: The ICE Study: Perceptions of E-Cigarettes and Synthetic Cooling Agents (R01)
Brief Title: Perceptions of E-Cigarettes and Synthetic Cooling Agents, the ICE Study
Acronym: ICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alayna Tackett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: OSU-23040; NCI-2023-06312 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA276696 (NIH)
Record Dates: First submitted 2023-11-30; First posted 2024-01-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Abuse Tobacco; Exposure
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Behavior Therapy; Specimen Handling

STUDY DESIGN:
Intervention Model Description: Randomization to condition order will be completed prior to study Visit 1. Each participant will receive a randomized ordering developed using a random sequence generator. Participants and data collection staff will be blinded to the order/conditions administered at each trial. The sequence list and subsequent participant ID numbers will be kept separate from data collection staff and will only be accessible by staff who will not be interacting with participants.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and study staff will be blinded to the study conditions delivered at each visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fruit flavored e-cigarette with synthetic cooling agents added (Active Comparator): Synthetic cooling agents will be added to fruit flavored e-liquid for this condition.
  Interventions: Behavioral: Behavioral Intervention; Other: Biospecimen Collection; Other: Survey Administration
- Fruit flavored e-cigarette (Active Comparator): Fruit flavored e-liquid will be used for this condition.
  Interventions: Behavioral: Behavioral Intervention; Other: Biospecimen Collection; Other: Survey Administration
- Tobacco flavored e-cigarette with synthetic cooling agents added (Active Comparator): Synthetic cooling agents will be added to tobacco flavored e-liquid for this condition.
  Interventions: Behavioral: Behavioral Intervention; Other: Biospecimen Collection; Other: Survey Administration
- Tobacco flavored e-cigarette (Active Comparator): Tobacco flavored e-liquid will be used for this condition.
  Interventions: Behavioral: Behavioral Intervention; Other: Biospecimen Collection; Other: Survey Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Receive and use flavored e-cigarettes (EC) as directed
Other: Biospecimen Collection — Undergo biosample sample collection
  Other Names: Biological Sample Collection; Specimen Collection
Other: Survey Administration — Complete surveys

SUMMARY:
This study evaluates how synthetic cooling additives like WS-3 and WS-23 impact e-cigarette perceptions, use behavior, and toxicant exposure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the abuse liability of e-liquids with and without the presence of synthetic cooling agents.

II. Determine the impact of synthetic cooling agents and flavor on EC puffing behavior (topography).

III. Determine the exposure ranges (harmful and potentially harmful constituents [HPHCs], other toxicants) from vaping e-liquids with and without the presence of synthetic cooling agents.

OUTLINE:

Participants attend 4 sessions where they receive 1 of 4 randomly assigned flavored e-cigarettes. Participants use the e cigarettes for vaping followed by ad libitum vaping. Participants also complete surveys and undergo biosample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-29 years
* Current exclusive e-cigarette (EC) user (defined as ≥ weekly use over the past 3 months)
* Willing to provide informed consent and abstain from using their EC at least 12 hours prior to the four lab sessions
* Read and speak English

Exclusion Criteria:

* Recently COVID-19+ (defined as positive test in the past 30 days) or a recent COVID-19 hospitalization (defined as a hospitalization within the past 6 months)
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* History of cardiac event or distress within the past 3 months
* Are currently pregnant, planning to become pregnant, or breastfeeding (will be verified with urine pregnancy test)
* Have suffered from any serious lung disease or infection (e.g. , tuberculosis, cystic fibrosis, or lung cancer) in the past 30 days
* Have hemophilia or another type of bleeding disorder
* Are blind, severely visually impaired, deaf, hard of hearing, or have a severe motor disability

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Satisfaction and psychological reward | Minute 5 of vaping session, Minute 35 of vaping session
  Satisfaction and psychological reward of e-cigarette (EC) vaping will be measured by the Modified Cigarette Evaluation Questionnaire (mCEQ). The mCEQ asks questions relating to satisfaction of using e-cigarettes on a scale from 0 (Not at all) - 6 (Extremely).
Sensory perceptions of EC vaping experience | Pre-vaping session
  Sensory perceptions of EC vaping will be measured by the Sensory E-cigarette Expectancies Scale (SEES) questionnaire. The SEES asks questions about sensory experiences associated with vaping on a scale from 0 (Never) - 4 (Almost Always).
E-cigarette puff topography | 35 Minute Vaping session
  Will be measured with a topography device that records frequency, duration, and flow rate of EC puffs. These measures are combined to inform overall EC puff behavior.
Levels of HPHC and other toxicant exposure from vaping e-liquids | After completion of sessions, estimated 4 years
  Topography data collected for all participants for each of the conditions vaped will be averaged to produce four human-derived puffing regimens. Machine vaping will be conducted for each of the four e-liquids using the associated human-derived puffing regimens to determine the range of HPHCs and other toxicants in mainstream EC vapor.
Appeal and Sensory | Minute 5 of vaping session, Minute 35 of vaping session
  Participants will rate appeal (e.g., liking, disliking) and sensory attributes (e.g., harshness, coolness) outcomes on Visual Analogue Scales (range, 0-100).

SECONDARY OUTCOMES:
Economic demand breakpoint | Minute 35 of vaping session
  The price point at which a participant is no longer willing to pay for a puff of the study e-liquid will be determined by an EC purchase task questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Alayna P Tackett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu